CLINICAL TRIAL: NCT00752713
Title: Strain-Encoded Magnetic Resonance Imaging for Evaluation of Left Ventricular Function and Acute Myocardial Infarction
Brief Title: Strain-Encoded Magnetic Resonance Imaging in Acute Myocardial Infarction
Acronym: 137-2005
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Mirja Neizel, MD, Medical Clinic III, University Hospital Heidelberg
Other Study IDs: SENC in AMI
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Acute Myocardial Infarction
Keywords: AMI,; Reperfusion; successful

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients presenting to hospital with AMI
  Interventions: Procedure: cardiac MRI
- 2: healthy volunteers as control group
  Interventions: Procedure: cardiac MRI

INTERVENTIONS:
Procedure: cardiac MRI — cardiac MRI at one time point for group 1 after intervention for group 2 at any time point
  Other Names: cardiac resonance magnetic imaging

SUMMARY:
The aim of the study was therefore to evaluate whether myocardial deformation imaging performed by SENC allows for quantification of regional left ventricular function and is related to transmurality states of infarcted tissue in patients with acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
CMR was performed in 38 consecutive patients with AMI 3±1 days after successful reperfusion using a clinical 1.5 Tesla MR-scanner. Ten healthy volunteers served as controls. SENC is a technique that directly measures peak circumferential strain from long-axis views and peak longitudinal strain from short axis views. Measurements were obtained for each segment in a modified 17 segment model. Wall motion and infarcted tissue were evaluated semi-quantitatively from SSFP cine sequences and contrast-enhanced-MR-images and were then related to myocardial strain. Comparison of peak circumferential strain assessed by SENC and MR-tagging was performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AMI after successful reperfusion
* Healthy volunteers in control group

Exclusion Criteria:

* No reperfusion

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Consecutive Patients with AMI 3+/-1 days after successful reperfusion
  * Ten healthy volunteers serving as control group
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Left ventricular function | 01.01.2007 until 01.02.2007

SECONDARY OUTCOMES:
Transmurality | 01.01.2007 until 01.02.2007

CONTACTS AND LOCATIONS:
Overall Officials: Mirja Neizel, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Neizel M, Korosoglou G, Lossnitzer D, Kuhl H, Hoffmann R, Ocklenburg C, Giannitsis E, Osman NF, Katus HA, Steen H. Impact of systolic and diastolic deformation indexes assessed by strain-encoded imaging to predict persistent severe myocardial dysfunction in patients after acute myocardial infarction at follow-up. J Am Coll Cardiol. 2010 Sep 21;56(13):1056-62. doi: 10.1016/j.jacc.2010.02.070. PMID 20846606